CLINICAL TRIAL: NCT06289907
Title: Effect of BH-HF3.0 on Vasomotor Symptoms (VMS) in Menopausal Women: A De-Centralized, Randomized, Double-Blinded, Placebo-Controlled Clinical Trial
Brief Title: Hot Flash and Night Sweat Virtual Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bonafide Health (Industry)
Collaborators: Lindus Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LH-BH-ADV-01
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-06

CONDITIONS: Menopause
Keywords: Menopause; Hot Flashes; Night Sweats
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Intervention Model Description: Decentralized, double-blind, placebo-controlled, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Active Comparator): Dietary supplement containing a proprietary botanical blend with NK3R antagonistic activity
  Interventions: Dietary Supplement: Bonafide-HF3.0
- Placebo group (Placebo Comparator): Placebo capsule containing:
  * Microcrystalline cellulose
  * Silicon dioxide micronized
  * Magnesium stearate
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bonafide-HF3.0 — Take 2 capsules once daily in the mornings with food
  Arms: Active group
Dietary Supplement: Placebo — Take 2 capsules once daily in the mornings with food
  Arms: Placebo group

SUMMARY:
The purpose of this research study is to evaluate the effectiveness of the study product on vasomotor symptoms (VMS) and overall menopause symptoms in healthy women, who are perimenopausal or postmenopausal, and aged 40 - 65.

DETAILED DESCRIPTION:
Menopause is characterized by the cessation of menstruation for 12 consecutive months. It is a natural phase in which a women's menstrual cycles permanently cease, with the transition often beginning around 51 years of age or older. Although menopause can be induced through procedures such as bilateral oophorectomy with or without hysterectomy and other medications, it most commonly occurs with the natural loss and depletion of ovarian follicles through aging. Common symptoms of menopause include changes in vaginal health and sexuality, loss of bladder control, changes in mood, decreased sleep quality, changes in body composition, and vasomotor symptoms (VMS).

Vasomotor symptoms (VMS), which include hot flashes and night sweats, occur in women at or around the time of menopause. Most women will experience these symptoms during the years surrounding their final menstrual period; however, there are some women that report VMS that persist for decades. The pathogenesis of VMS has not been fully understood, but the pathways involving estrogen, norepinephrine, and serotonin are hypothesized to cause altered homeostatic thermoregulatory mechanisms. VMS can have a negative impact on quality of life by disrupting both sleep and mood.4 About one-third of women in the United States are older than 50 years of age, the typical age of onset. Approximately 75% of women in this age group (i.e., 40 to 50 million currently) will experience hot flashes.

Treatments for VMS range significantly from prescription medications to over-the-counter therapies (non-prescription) to lifestyle modifications. Hormone replacement therapy (HRT) still remains the most common and effective treatment. Hormone replacement therapy, using estrogen or estrogen-progestin-containing products, reduces the frequency and severity of hot flashes by 75-79%. Although hormone replacement therapy is generally well tolerated, it has been linked to an increased risk of breast cancer. Due to this concern, it is recommended to use hormone replacement therapy for the shortest duration and lowest dose possible, based on individual circumstances and needs. Additionally, many healthcare practitioners and patients seek alternative solutions to HRT for personal and medical reasons. Alternatives to HRT vary from hypnosis and dietary supplements, including vitamin E, black cohosh, and phytoestrogens, all which drastically differ in their VMS mitigation effectiveness. There is a need for an effective and safe treatment of VMS for menopausal women, and dietary supplements may fill this role.

The SP for this study is Bonafide Health's Bonafide-HF3.0. Bonafide-HF3.0 contains green tea extract (GTE), curcumin, and phycocyanin sourced from Spirulina "Blue-Green" algae.

This double-blind placebo-controlled (DBPC) study will be conducted to evaluate the effectiveness of Bonafide-HF3.0 on vasomotor symptoms and overall menopausal symptoms in healthy women, aged 40-65, who are perimenopausal and menopausal.

ELIGIBILITY:
Inclusion Criteria

* Healthy women who are 40 to 65 years of age (inclusive).
* Have a body mass index (BMI) between 18.5 to 34.9 kg/m2 (inclusive).
* Have self-reported menopausal symptoms for the past 6 months (perimenopause, post-menopause).
* Have self-reported at least 5 moderate to severe vasomotor symptoms (hot flashes and/or night sweats) most days of the week.
* In good general health (no active or uncontrolled diseases or conditions) and able to consume the study product.
* Agree to refrain from treatments listed in the concomitant meds section within the defined timeframe.
* Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria

* Individuals who are lactating, pregnant, or planning to become pregnant during the study.
* Currently incarcerated prisoners
* Use of any treatment for menopausal symptoms or other concomitant treatments listed in Section 11.4.
* Have a known sensitivity, intolerability, or allergy to any of the study product or their excipients.
* Received a vaccine for COVID-19 in the two weeks prior to screening or planning to receive during the study period, current COVID-19 infections, or currently have the post COVID-19 condition as defined by World Health Organization (WHO) (i.e., individuals with a history of probable or confirmed SARS-CoV-2 infection, usually three months from the onset of COVID-19 with symptoms that last for at least two months and cannot be explained by an alternative diagnosis).
* Have a positive medical history of heart disease, renal disease, hepatic impairment, or active systemic infection (i.e., Lyme disease, TB, HIV).
* History of cancer (except localized skin cancer without metastases) within 1 year prior to screening.
* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential subject at risk because of participation in the study or influence the results or the potential subject's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs (i.e., Crohn's disease, short bowel, acute or chronic pancreatitis, gastric bypass procedures, or pancreatic insufficiency).
* Active vaginal infections/abnormalities (e.g., active urinary tract infection (UTI), genital hemorrhage of unknown origin, pelvic inflammatory disease (PID)). Note: screened participants with infections would be eligible to participate two weeks after completing their treatment/antibiotics (wash-out period).
* Participant has an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea).
* Major surgery in three months prior to screening or planned major surgery during the study.
* History of alcohol or substance abuse in the last 3 years.
* Use of any vaginal medications, rinses, or moisturizers, or other items including cooling devices, cooling mattresses, cooling sprays, or patches purposed for hot flash control (i.e., V-qool patch, estrogen cream, etc.) one week before and during study.
* Participation in another clinical or research trial.
* Any other active or unstable medical conditions or use of medications/supplements/ therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy women, who are perimenopausal or postmenopausal, and aged 40 - 65.
Enrollment: 80 (Estimated)
Dates: Start 2023-07-09 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
To determine the effects of the Study Product (SP) compared to placebo on hot flash symptoms | 12 weeks
  The number and severity of hot flashes assessed via participant diary tracking (electronic)
To determine the effects of the SP compared to placebo on hot flash symptoms | 12 weeks
  The number and severity of night sweats assessed via participant diary tracking (electronic)
To determine the effects of the SP compared to placebo on hot flash symptoms | 12 weeks
  Change from baseline for the Hot Flash Related Daily Interference Scale (HFRDIS) scores at EOS
To determine the effects of the SP compared to placebo on vasomotor symptoms | 12 weeks
  Change from baseline for the Visual Analog Scale (VAS) Vasomotor Symptoms Questionnaire at EOS
To determine the effects of the SP compared to placebo on overall menopausal symptoms | 12 weeks
  Change from baseline for the Menopausal Rating Scale (MRS) in scores at EOS
To determine the effects of the SP compared to placebo on overall menopausal symptoms | 12 weeks
  Change from baseline for the Visual Analog Scale (VAS) Menopausal Symptoms Questionnaire in scores at EOS
To determine the effects of the SP compared to placebo on quality of life | 12 weeks
  Change from baseline in Menopause-Specific Quality of Life (MENQOL) scores

CONTACTS AND LOCATIONS:
Overall Officials: Trisha VanDusseldorp, Ph.D., Study Director — Bonafide Health, LLC
Locations (1):
- Lindus Health, Inc., London, United Kingdom

IPD SHARING:
Plan to Share IPD: No